CLINICAL TRIAL: NCT03510572
Title: Clinical Evaluation of [18F]PI-2620 Positron Emission Computed Tomography for Imaging Tau Protein in Patients With Tauopathies and Healthy Volunteers: Phase 0 Study
Brief Title: Evaluation of [18F]PI-2620 as a Potential Positron Emission Computed Tomography Radioligand for Imaging Tau Protein in the Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jae Seung Kim, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI-18001
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Healthy Volunteer; Alzheimer Disease; Frontotemporal Dementia; Parkinson Disease
Keywords: [18F]PI-2620, tauopathy, positron emission computed tomography
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Parkinson Disease; Tauopathies | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteer (Experimental): Cognitively healthy subjects will receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620
- Alzheimer's Disease (Experimental): Alzheimer's Disease Subjects will receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620
- Frontotemporal dementia (Experimental): frontotemporal dementia Subjects will receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620
- Parkinson's disease (Experimental): Parkinson's disease Subjects will receive a single IV injection of [18F]PI-2620.
  Interventions: Drug: [18F]PI-2620

INTERVENTIONS:
Drug: [18F]PI-2620 — Imaging for evaluating the accumulation of abnormal tau protein in the brain
  Other Names: FluoroTau

SUMMARY:
The overall goal of this imaging trial is to evaluate [18F]PI-2620, a tau targeted positron emission computed tomography radioligand, in individuals with tauopathies and healthy volunteers (HV).

ELIGIBILITY:
Inclusion Criteria:

1. General Subject Inclusion Criteria

   In order to be eligible for participation in this trial, the subject must:
   * Be ≥ 40 and < 80 years of age at the Screening Visit.
   * Be able to read at a 6th grade level or equivalent, (as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation.)
   * Be able to speak, read, hear, and understand the language of the trial staff, and the informed consent form, and possess the ability to respond verbally to questions, follow instructions, and complete questionnaires and detailed neuropsychological test.
   * Have results of clinical laboratory tests/physical examination, vital signs, and ECG within normal limits (at 90 days prior to [18F]PI-2620 positron emission computed tomography) or clinically acceptable to the investigator at screening.
   * If female, not be of childbearing potential as indicated by one of the following
   * Each subject (or legal representative) must sign the informed consent form in accordance with local requirements after the scope and nature of the investigation have been explained to them, and before screening assessments.
2. Cognitively Healthy Subjects
3. Subjects with Alzheimer's disease
4. Subjects with frontotemporal dementia
5. Subjects with Parkinson's disease

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject fulfil any single criteria described below:

1. General Exclusion Criteria

   * Based on the investigators' judgement, if the patient is not capable of communicating with the site personnel, if the patient is not proficient in the language in which the psychometric tests will be completed, or if the patient is not sufficient for compliance with the study procedures.
   * The patient has an abnormal physical examination or abnormal laboratory test results at the screening that are clinically significant to affect results of the research, as judged by the investigator.
   * If the patient has or is suspicious of having a hypersensitivity or allergy to [18F] PI-2620 or its derivatives.
   * The patient is pregnant, is attempting to become pregnant, or is nursing (breast-feeding) children.
   * The patient has a history of alcoholism or drug dependency/abuse within the last 2 years before screening.
   * The patient has contraindications to undergo positron emission computed tomography or MRI, which include but are not restricted to the examples below: claustrophobia, cardiac pacemaker, metal devices around the eye or spinal cord, cochlear implant, etc.) at the screening visit.
   * The patient has been treated with any investigational medicinal product (IMP) within 30 days prior to the screening visit.
2. Cognitively Healthy Subjects
3. Subjects with Alzheimer's disease
4. Subjects with frontotemporal dementia
5. Subjects with Parkinson's disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Cross-sectional [18F]PI-2620 Imaging Results | 60-90 minutes post injection
  Compare Standard uptake value ratio (SUVR) and distribution of [18F]PI-2620 in subjects with tauopathies and cognitively healthy individuals.
.Assess the rate of change of tau deposition as measured by [18F]PI-2620 uptake (SUVR) over time | 60-90 minutes post injection
  Compare Standard uptake value ratio (SUVR) and distribution of [18F]PI-2620 in subjects with tauopathies and cognitively healthy individuals.

SECONDARY OUTCOMES:
Correlation between standard uptake value ratio (SUVR) of [18F]PI-2620 positron emission computed tomography and neuropsychiatric test scores | 60-90 minutes post injection
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]PI-2620 positron emission computed tomography and scores of neuropsychiatric test
Correlation between standard uptake value ratio (SUVR) of [18F]PI-2620 positron emission computed tomography and indices of structural MRI | 60-90 minutes post injection
  We will evaluate correlation between standard uptake value ratio (SUVR) [18F]PI-2620 positron emission computed tomography and indices of structural MRI including cortical thickness, hippocampal atrophy.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided